CLINICAL TRIAL: NCT05620641
Title: Comparative Clinical Study Among Ondansetron and Gabapentin in Preventing Postoperative Nausea and Vomiting After Laparoscopic Sleeve Gastrectomy
Brief Title: Ondansetron and Gabapentin in Preventing Postoperative Nausea and Vomiting After Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Gamal Moussa, Assistant Lecturer at Clinical Pharmacy department , Faculty of Pharmacy -Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 35647
Record Dates: First submitted 2022-11-11; First posted 2022-11-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Post Operative Nausea and Vomiting; Sleeve Gastrectomy; Morbid Obesity
Keywords: Postoperative Nausea and Vomiting; Laparoscopic Sleeve Gastrectomy; ondansetron; gabapentine
MeSH Terms: conditions — Vomiting; Obesity, Morbid; Postoperative Nausea and Vomiting | interventions — Ondansetron; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): include 50 patients scheduled for sleeve gastrectomy
  Interventions: Drug: Ondansetron 8mg
- Group 2 (Experimental): include 50 patients scheduled for sleeve gastrectomy
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Ondansetron 8mg — 50 patients will receive intravenous ondansetron 8 mg before the end of surgery.
  Other Names: zofran
  Arms: Group 1
Drug: Gabapentin — 50 patients will receive 600 mg oral gabapentin 1 h before anesthesia.
  Arms: Group 2

SUMMARY:
The aim of this study is to compare the possible efficacy of ondansetron and gabapentin on postoperative nausea and vomiting in patient with morbid obesity who will undergo laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
This study will be a double blind randomized, controlled, parallel, study. A total of1 00 morbidly obese patients who will be scheduled for sleeve gastrectomy will be included in the study. The patients will be selected from those attending Gastrointestinal and Laparoscopic Surgery Unit, General Surgery Department, Tanta University Hospital, Tanta, Egypt. The participants will be randomized into two groups by closed envelop method,

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients will be included.
* Morbidly obese patients scheduled for sleeve gastrectomy with BMI ≥35 kg/m2 with the presence of comorbidity such as hypertension, arthritis, and diabetes.
* Morbidly obese patients scheduled for sleeve gastrectomy with BMI ≥ 40 kg/m2 without comorbidity.
* Patients fit for anesthesia and surgery.

Exclusion Criteria:

* - Patients with BMI >55 kg/m2.
* Patients with previous procedures for the treatment of obesity.
* Pregnant females and lactating women.
* Patients with psychological or psychiatric disease
* Administration of antiemetic medication or systemic corticosteroids within 24 hours before surgery
* Patients who experienced vomiting within 24 hours before surgery.
* Patients with history of alcohol or drug abuse.
* Patients with hypersensitivity or contraindications to any of the drugs used in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study will be the complete response within the first 48 h after surgery. | The first 48 hours after surgery.
  Complete response is defined as the absence of PONV and the lack of a need for rescue antiemetic therapy

SECONDARY OUTCOMES:
change in the level of the biological parameter vasopressin | The first 48 hours after surgery.
  5 ml of venous blood will be withdrawn from each participant by antecubital venipuncture. Blood samples will be centrifuged at 3000 rpm for 15 min to separate sera. Sera will be kept at deep freeze (-80°C) until analysis of serum concentrations of vasopressin
change in the level of the biological parameter dopamine | The first 48 hours after surgery.
  5 ml of venous blood will be withdrawn from each participant by antecubital venipuncture. Blood samples will be centrifuged at 3000 rpm for 15 min to separate sera. Sera will be kept at deep freeze (-80°C) until analysis of serum concentrations of dopamine
change in the level of the biological parameter substance p | The first 48 hours after surgery.
  5 ml of venous blood will be withdrawn from each participant by antecubital venipuncture. Blood samples will be centrifuged at 3000 rpm for 15 min to separate sera. Sera will be kept at deep freeze (-80°C) until analysis of serum concentrations of substance p
change in the level of the biological parameter Serotonin | The first 48 hours after surgery.
  5 ml of venous blood will be withdrawn from each participant by antecubital venipuncture. Blood samples will be centrifuged at 3000 rpm for 15 min to separate sera. Sera will be kept at deep freeze (-80°C) until analysis of serum concentrations of Serotonin
change in the level of the biological parameter Tachykinin 1 | The first 48 hours after surgery.
  5 ml of venous blood will be withdrawn from each participant by antecubital venipuncture. Blood samples will be centrifuged at 3000 rpm for 15 min to separate sera. Sera will be kept at deep freeze (-80°C) until analysis of serum concentrations of Tachykinin 1

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrointestinal and Laparoscopic Surgery Unit, General Surgery Department, Tanta University Hospital, Tanta, Egypt, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No